CLINICAL TRIAL: NCT01859936
Title: Randomized Multicenter Trial Assessing if Preoperative MRI Breast in Women Under 56 Years With Breast Cancer Will Change Primary Treatment
Brief Title: Will Preoperative MRI Breast in Women Under 56 Years With Breast Cancer Change Primary Treatment
Acronym: POMB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Brita Arver, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: POMB
Record Dates: First submitted 2013-05-16; First posted 2013-05-22 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preoperative breast MRI (Experimental): The intervention is that preoperative MRI breast will be performed in women under 56 years with newly diagnosed breast cancer
  Interventions: Device: MRI
- no MRI breast (No Intervention): The arm type description implies that no MRI breast will be performed to women under 56 years with newly diagnosed breast cancer

INTERVENTIONS:
Device: MRI — The intervention is that preoperative MRI breast will be performed in 220 women under 56 years with newly diagnosed breast cancer. Aims are to analyze if the intervention will affect primary management, decrease the number of reoperations and to analyze if the intervention leads to an increasing number of unnecessary mastectomies compared to the non intervention arm.
  Arms: preoperative breast MRI

SUMMARY:
The study is a prospective randomised multicenter trial assessing the additional value of breast MRI in women under 56 years of age with newly diagnosed breast cancer. Will preoperative breast MRI change treatment regimen? Will preoperative breast MRI reduce the number of primary surgeries? Will preoperative breast MRI increase the rate of mastectomies? Will preoperative breast MRI be cost effective?

DETAILED DESCRIPTION:
Completed: the study has concluded normally; participants are no longer being examined or treated (i.e., last patient's last visit has occurred)

ELIGIBILITY:
Inclusion Criteria:

* Women under 56 years of age
* Newly diagnosed breast cancer
* Swedish or English speaking

Exclusion Criteria:

* Claustrophobia
* Pregnancy
* Renal failure
* Metal items in patients

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change of treatment plan | 14 days
  Did breast magnetic resonance imaging add information about the tumour that changed primary treatment plan

SECONDARY OUTCOMES:
Did breast magnetic resonance imaging reduce the number of reoperation during primary management | 6 months
Did breast magnetic resonance imaging increase the number of mastectomies | 6 months
Did breast magnetic resonance imaging affect cost | 6 months

OTHER OUTCOMES:
Is the sensitivity of breast MRI dependant on density and/or on age | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Brita Arver, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska Univeristy Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Gonzalez V, Arver B, Lofgren L, Bergkvist L, Sandelin K, Eriksson S. Impact of preoperative breast MRI on 10-year survival of patients included in the Swedish randomized multicentre POMB trial. BJS Open. 2021 Sep 6;5(5):zrab088. doi: 10.1093/bjsopen/zrab088. PMID 34611701